CLINICAL TRIAL: NCT03326141
Title: Community-based Intervention Effects on Older Adults' Physical Activity and Falls (R01)
Brief Title: Community-based Intervention Effects on Older Adults' Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1607S90922; 1R01NR016705-01A1 (NIH)
Record Dates: First submitted 2017-09-01; First posted 2017-10-31 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Exercise; Physical Activity; Accidental Fall; Motivation; Older Adults
MeSH Terms: conditions — Motor Activity | interventions — Health

STUDY DESIGN:
Intervention Model Description: Our research team will conduct a 2 x 2 factorial experiment testing the individual and combined effects of two empirically and theoretically relevant sets of behavior change strategies on community-dwelling older adults' physical activity.
Who Masked: Outcomes Assessor
Masking Description: The specific content of the intervention condition/arm that is assigned to each participant will be masked from data collectors/outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Otago+PAM+Health / Wellness topics (Active Comparator): Condition 1:
  Otago Exercise Program adapted for delivery to small groups; a physical activity monitor such as a Fitbit (PAM); and, information about health and wellness (8) topics guided by content in the National Institute on Aging (NIA) and Centers for Disease Control and Prevention websites.
  Interventions: Behavioral: Otago Exercise Program; Device: Physical activity monitors (e.g., Fitbit); Other: Information about Health and Wellness
- Otago + PAM + Interpersonal strategies (Experimental): Condition 2:
  Otago Exercise Program adapted for delivery to small groups; a PAM (e.g.,Fitbit); 5 Interpersonal behavior change strategies; and, information about health and wellness topics (1) guided by content in the National Institute on Aging (NIA) and Centers for Disease Control and Prevention websites.
  Interventions: Behavioral: Otago Exercise Program; Device: Physical activity monitors (e.g., Fitbit); Behavioral: Interpersonal Behavior Change Strategies
- Otago, PAM, Intrapersonal strategies (Experimental): Condition 3:
  Otago Exercise Program adapted for delivery to small groups; a PAM (e.g.,Fitbit); 5 Intrapersonal behavior change strategies; and, health and wellness topics (1) guided by content in the National Institute on Aging (NIA) and Centers for Disease Control and Prevention websites.
  Interventions: Behavioral: Otago Exercise Program; Device: Physical activity monitors (e.g., Fitbit); Behavioral: Intrapersonal Behavior Change Strategies
- Otago,PAM, Inter+Intra strategies (Experimental): Condition 4:
  Otago Exercise Program adapted for delivery to small groups; a PAM (e.g., Fitbit); 5 Interpersonal behavior change strategies; and, 5 Intrapersonal behavior change strategies
  Interventions: Behavioral: Otago Exercise Program; Device: Physical activity monitors (e.g., Fitbit); Behavioral: Interpersonal Behavior Change Strategies; Behavioral: Intrapersonal Behavior Change Strategies

INTERVENTIONS:
Behavioral: Otago Exercise Program — The program has been adapted for groups and includes 5 flexibility movements (e.g., back extension and ankle, head, neck, trunk movements), 5 leg strengthening exercises (knee extensor, knee flexor, hip abductor, ankle plantar flexes, ankle dorsiflexes), 12 balance movements (knee bends, backwards walking, walking and turning, sideways walking, tandem stance, tandem walk, one leg stand, heel walking, toe walking, heel-toe walking backwards, sit to stand, stair walking), and a walking plan. The number, intensity and duration of movements are individualized according to preference and ability and they are gradually progressed.
Device: Physical activity monitors (e.g., Fitbit) — We will use Fitbit Charge 2 (or an equivalent). Features essential for this research include built-in accelerometers that accurately measure steps and physical activity (PA) duration.Participants will have a brief orientation to these during baseline data collection and have the opportunity to return demonstrate. In addition, RAs will be available to help participants troubleshoot, as needed, via telephone and in person, after intervention meetings. Intervention meetings include discussions about the PAMs, but topics vary according to assigned study condition.
  Other Names: PAM
Behavioral: Interpersonal Behavior Change Strategies — The interpersonal content will include facilitated discussed about including PA into social routines, identifying and problem-solving social and environmental barriers to PA, social support for exercise, and friendly social comparisons about practicing PA outside the small group setting and interpreting/ sharing data.
  Arms: Otago + PAM + Interpersonal strategies; Otago,PAM, Inter+Intra strategies
Behavioral: Intrapersonal Behavior Change Strategies — The intrapersonal content will include encouragement and guidance to identify baseline PA patterns, develop and refine personally meaningful goals and plans, identify and problem solve personal barriers to staying physically active, integrate PA into personal routines, and monitor goal outcomes
  Arms: Otago, PAM, Intrapersonal strategies; Otago,PAM, Inter+Intra strategies
Other: Information about Health and Wellness — Information about health and wellness varies in dose, according to time spent in each condition that addresses behavior change. Topics in condition 1 include sleep, vaccinations, supplements, fall risk factors, memory, hearing and pain guided by information for older adults available on the NIA and CDC websites. Topics in conditions 2 and 3 include fall risk factors and sleep. Topics in condition 4 include fall risk factors.
  Arms: Otago+PAM+Health / Wellness topics

SUMMARY:
The research team will conduct a 2 x 2 factorial experiment testing the individual and combined effects of two empirically and theoretically relevant sets of behavior change strategies on community-dwelling older adults' physical activity. To do this the investigators will randomize participants >= 70 years old (n = 308) to 1 of 4 experimental conditions. All conditions include an evidence-based physical activity protocol endorsed by Centers for Disease Control and Prevention (CDC) for use by all older adults, including those with frailty and multiple co-morbidities and the commercially available physical activity monitor (e.g., Fitbit) to augment intervention delivery. Intervention components that are experimental and vary by condition are the sets of behavior change strategies which will be combined with the physical activity protocol and the physical activity monitor. Condition 1 has no specific behavior change strategies; Condition 2 includes an intervention component comprised of 5 interpersonal behavior change strategies, such as facilitating social support and social comparison; Condition 3 includes an intervention component comprised of 5 intrapersonal behavior change strategies, such as setting personally meaningful goals; and Condition 4 includes both sets of behavior change strategies -- 5 interpersonal strategies combined with 5 intrapersonal behavior change strategies.

DETAILED DESCRIPTION:
To fully examine the effects of these experimental components, The investigators have delineated Primary, Secondary and Exploratory Aims:

Primary Aim: Determine which experimental intervention component(s) increase PA among community-dwelling older adults post-intervention: immediately, 6 months, and 12 months. Hypothesis: Participants receiving the interpersonal set of behavior change strategies (conditions 2 and 4) will have clinically meaningful increases in PA post- intervention (at all 3 time-points), compared to participants not receiving these strategies (conditions 1 and 3).

Secondary Aim: Determine which experimental intervention component(s)decrease fall occurrence and increase quality of life (QOL) among community-dwelling older adults 12 months post-intervention. Hypotheses: Participants receiving the set of interpersonal behavior change strategies will have clinically meaningful reductions in falls and increases in QOL, 12 months post-intervention, compared to participants not receiving these strategies.

Exploratory Aim: Evaluate experimental intervention component effects on targeted psychosocial constructs (social support; readiness; self-regulation) and physical constructs (functional leg strength and balance), which are theorized as mechanisms of change--and whether these mechanisms mediate the effects of experimental intervention components on PA and falls. Hypotheses: Receiving the interpersonal behavioral change strategies, relative to not receiving these strategies, will elicit increases in targeted psychosocial constructs and increases in physical constructs, which in turn will mediate the intervention's effects on PA behavior and falls.

ELIGIBILITY:
Inclusion Criteria:

* ≥70 years of age
* English speaking
* Low levels of PA (below recommended guidelines)
* Self-reported fall risk as guided by the CDC, Steadi fall risk screener

  * One or more falls in the last year
  * Unsteadiness when standing or walking
  * Worries about falling
* Participants who self-report the following symptoms will require clearance from a primary provider (as guided by the Exercise and Screening for You Questionnaire)

  * Pain, tightness or pressure in chest during PA (walking, climbing stairs, household chores, similar activities) that have not been checked and/ or treated by a healthcare provider
  * Current dizziness that have not been checked and/ or treated by a healthcare provider
  * Current, frequent falls that have not been checked and/ or treated by a healthcare provider

Exclusion Criteria:

* Lower extremity injury or surgery within the past 6 weeks
* Inability to walk
* Formal diagnosis of neurocognitive impairment or dementia

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 309 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siobhan K McMahon, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota - School of Nursing, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this study, including baseline characteristics and outcome variables, will be shared via Data Repository at the University of Minnesota after March 2024
Supporting Information: Study Protocol, ICF
Time Frame: November 17, 2017 to September 2, 2022
Access Criteria: IRB approval

REFERENCES:
- [Derived] McMahon SK, Lewis BA, Guan W, Wang Q, Hayes SM, Wyman JF, Rothman AJ. Effect of Intrapersonal and Interpersonal Behavior Change Strategies on Physical Activity Among Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2024 Feb 5;7(2):e240298. doi: 10.1001/jamanetworkopen.2024.0298. PMID 38421648

RESULTS

PARTICIPANT FLOW:
Groups:
- Otago+PAM+Health / Wellness Topics: Condition 1:
  Otago Exercise Program (OEP) adapted for delivery to small groups. In total, this protocol includes 5 flexibility movements, 5 leg-strengthening movements, and 12 balance-challenging movements. The number intensity and duration (dosages) are individualized according to preference and ability. OEP movements are gradually progressed across the 8-week intervention. A physical activity monitor (PAM) (Fitbit Charge 2) with initial orientation and ongoing support.
  Health and wellness information (attention control content) guided by content in the National Instituteon Aging (NIA) and Centers for Disease Control and Prevention websites.
- Otago + PAM + Interpersonal Strategies: Condition 2:
  1. Otago Exercise Program (OEP) adapted for delivery to small groups. In total, this protocol includes 5 flexibility movements, 5 leg-strengthening movements, and 12 balance-challenging movements. The number intensity and duration (dosages) are individualized according to preference and ability. OEP movements are gradually progressed across the 8-week intervention.
  2. A physical activity monitor (PAM) (Fitbit Charge 2) with initial orientation and ongoing support.
  3. Interpersonal behavior change strategies including peer-to-peer sharing and learning about using activities in everyday routines as prompts for movement, identifying and problem solving environmental barriers to physical activity, ways to increase social support for physical activity, and friendly social comparison of experiences performing OEP movements and home and other locations of choice, staying motivated to practice OEP movements long-term.
- Otago, PAM, Intrapersonal Strategies: Condition 3:
  1. Otago Exercise Program (OEP) adapted for delivery to small groups. In total, this protocol includes 5 flexibility movements, 5 leg-strengthening movements, and 12 balance-challenging movements. The number intensity and duration (dosages) are individualized according to preference and ability. OEP movements are gradually progressed across the 8-week intervention.
  2. A physical activity monitor (PAM) (Fitbit Charge 2) with initial orientation and ongoing support.
  3. Intrapersonal behavior change strategies including to develop physical activity related goals and action plans, self-assess goal attainment and action plan implementation-adjust accordingly, identify and problem solve personal barriers to physical activity, develop a habit of one or more OEP movements.
- Otago,PAM, Inter+Intra Strategies: Condition 4:
  1. Otago Exercise Program (OEP) adapted for delivery to small groups. In total, this protocol includes 5 flexibility movements, 5 leg-strengthening movements, and 12 balance-challenging movements. The number intensity and duration (dosages) are individualized according to preference and ability. OEP movements are gradually progressed across the 8-week intervention.
  2. A physical activity monitor (PAM) (Fitbit Charge 2) with initial orientation and ongoing support.
  3. Interpersonal behavior change strategies including peer-to-peer sharing and learning about using activities in everyday routines as prompts for movement, identifying and problem solving environmental barriers to physical activity, ways to increase social support for physical activity, and friendly social comparison of experiences performing OEP movements and home and other locations of choice, staying motivated to practice OEP movements long-term.
  4. Intrapersonal behavior change strategies including to develop physical activity related goals and action plans, self-assess goal attainment and action plan implementation-adjust accordingly, identify and problem solve personal barriers to physical activity, develop a habit of one or more OEP movements
Period: Overall Study
Arm/Group | Otago+PAM+Health / Wellness Topics | Otago + PAM + Interpersonal Strategies | Otago, PAM, Intrapersonal Strategies | Otago,PAM, Inter+Intra Strategies
Started | 78 | 78 | 76 | 77
Completed | 77 | 76 | 74 | 75
Not Completed | 1 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Otago+PAM+Health / Wellness Topics: Condition 1:
  1. Otago Exercise Program (OEP) adapted for delivery to small groups. In total, this protocol includes 5 flexibility movements, 5 leg-strengthening movements, and 12 balance-challenging movements. The number intensity and duration (dosages) are individualized according to preference and ability. OEP movements are gradually progressed across the 8-week intervention.
  2. A physical activity monitor (PAM) (Fitbit Charge 2) with initial orientation and ongoing support.
  3. Health and wellness information (attention control content) guided by content in the National Instituteon Aging (NIA) and Centers for Disease Control and Prevention websites.
- Total: Total of all reporting groups
Arm/Group | Otago+PAM+Health / Wellness Topics | Otago + PAM + Interpersonal Strategies | Otago, PAM, Intrapersonal Strategies | Otago,PAM, Inter+Intra Strategies | Total
Number analyzed (Participants) | 78 | 78 | 76 | 77 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.8 (5) | 77.7 (5) | 77.3 (5) | 76.6 (5.1) | 77.4 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 59 | 59 | 58 | 240
  Male | 14 | 19 | 17 | 19 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 10 | 16 | 9 | 48
  White | 65 | 66 | 57 | 67 | 255
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Quantity of Physical Activity Measured Objectively
Description: Average weekly minutes of total physical activity per week (light, moderate and vigorous intensities) as captured from PAM data (Fitbit Charge-2)
Time Frame: Baseline and Post-Intervention (one week, six months, twelve months)
Population: Number analyzed at baseline and post-intervention (one week, six months, twelve months) represent the number of participants in the study at that time. Numbers decrease across longitudinal time points due to participant withdrawal or loss to follow up
Measure: Mean (Standard Deviation); unit: minutes per day
Groups:
- Otago,PAM, Inter+Intra Strategies: Condition 4:
  1. Otago Exercise Program (OEP) adapted for delivery to small groups. In total, this protocol includes 5 flexibility movements, 5 leg-strengthening movements, and 12 balance-challenging movements. The number intensity and duration (dosages) are individualized according to preference and ability. OEP movements are gradually progressed across the 8-week intervention.
  2. A physical activity monitor (PAM) (Fitbit Charge 2) with initial orientation and ongoing support.
  3. Intrapersonal behavior change strategies including to develop physical activity related goals and action plans, self-assess goal attainment and action plan implementation-adjust accordingly, identify and problem solve personal barriers to physical activity, develop a habit of one or more OEP movements.
Arm/Group | Otago+PAM+Health / Wellness Topics | Otago + PAM + Interpersonal Strategies | Otago, PAM, Intrapersonal Strategies | Otago,PAM, Inter+Intra Strategies
Number analyzed (Participants) | 78 | 78 | 76 | 77
minutes per day
  Baseline | 177.9 (62.2) | 167.7 (79.1) | 185.9 (70.5) | 177.9 (72.7)
  one week post-intervention: number analyzed (Participants) | 77 | 77 | 75 | 76
  one week post-intervention | 180.5 (68.5) | 193.1 (82.1) | 181 (68.2) | 209.1 (79.2)
  six months post-intervention: number analyzed (Participants) | 77 | 77 | 75 | 75
  six months post-intervention | 180 (73.8) | 185.7 (84) | 175.1 (68.9) | 198 (78)
  twelve months post-intervention: number analyzed (Participants) | 77 | 76 | 74 | 75
  twelve months post-intervention | 174.3 (72.0) | 190.3 (99.1) | 167.7 (68.6) | 192.9 (80.4)

2. Primary Outcome: Physical Activity Scale for the Elderly (PASE)
Description: Self-report Measure of Physical Activity. PASE is a validated questionnaire to measure the amount of physical activity in people over the age of 65 including types (e.g., walking, recreational, exercise, housework, care-giving). Scores, accounting for frequency, duration and intensity of physical activity are calculated and typically range from 0 to 793, with higher value representing more physical activity.
Time Frame: Baseline and Post-Intervention (one week, six months, twelve months)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Total PASE Score
Arm/Group | Otago+PAM+Health / Wellness Topics | Otago + PAM + Interpersonal Strategies | Otago, PAM, Intrapersonal Strategies | Otago,PAM, Inter+Intra Strategies
Number analyzed (Participants) | 78 | 78 | 76 | 77
Total PASE Score
  Baseline | 102.2 (46.4) | 108.3 (66.6) | 110.6 (44) | 101.8 (48.5)
  One week post-intervention: number analyzed (Participants) | 77 | 77 | 75 | 76
  One week post-intervention | 111.1 (47.3) | 119.2 (69.9) | 120.7 (56.2) | 121.1 (58.7)
  Six months post-intervention: number analyzed (Participants) | 77 | 77 | 75 | 75
  Six months post-intervention | 106.7 (53.0) | 118.2 (65.1) | 119.5 (65.8) | 112.2 (60.1)
  Twelve months post-intervention: number analyzed (Participants) | 77 | 76 | 74 | 75
  Twelve months post-intervention | 107.1 (60.0) | 113.8 (66.8) | 123.0 (92.3) | 112.4 (60.9)

3. Secondary Outcome: Fall Rate
Description: Falls per person year, assessed via prospective monthly calendars
Time Frame: 12 months post intervention
Measure: Number; unit: Falls per person year
Arm/Group | Otago+PAM+Health / Wellness Topics | Otago + PAM + Interpersonal Strategies | Otago, PAM, Intrapersonal Strategies | Otago,PAM, Inter+Intra Strategies
Number analyzed (Participants) | 77 | 76 | 74 | 75
Falls per person year | 0.9 | 1.0 | 0.9 | 1.1

4. Secondary Outcome: Number of Participants With Moderate or Major Injuries From Falls
Description: Number of injuries from falls was measured via prospective falls calendars mailed to participants monthly with return addressed/stamped envelopes. Circumstances and injuries related to each fall were documented on the calendars. Calendar documentation each fall was verified and detailed through phone conversations between participants and trained research staff. Moderate and Major injuries from falls were categorized according to the Agency for Healthcare Research and Quality with moderate injuries defined as necessitating sutures, skin glue, splinting, and or involving muscle or joint strain. Major injuries were defined as those associated with internal injuries or a need for surgery, casting, traction, or neurological consults.
Time Frame: 12 months post intervention
Measure: Number; unit: Participants
Arm/Group | Otago+PAM+Health / Wellness Topics | Otago + PAM + Interpersonal Strategies | Otago, PAM, Intrapersonal Strategies | Otago,PAM, Inter+Intra Strategies
Number analyzed (Participants) | 77 | 76 | 74 | 75
Participants
  Number of moderate injurious falls | 6 | 7 | 6 | 6
  Number of major injurious falls | 1 | 2 | 2 | 1

5. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Scale v1.2 Global Health
Description: Using the Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Questionnaire 1.2. Two constructs from this questionnaire were converted to t scores: self-reported physical health and self-reported mental health. . Mean t scores are 50, which indicates the adult population mean with a standard deviation of 10. Higher t scores are considered better, or healthier, for self-reported physical health and mental health.
  No clinically relevant thresholds were described in this study.
Time Frame: Baseline and post-intervention: one-week, six months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Otago+PAM+Health / Wellness Topics | Otago + PAM + Interpersonal Strategies | Otago, PAM, Intrapersonal Strategies | Otago,PAM, Inter+Intra Strategies
Number analyzed (Participants) | 78 | 78 | 76 | 77
T score
  Physical Health: Baseline | 39.2 (4.9) | 39.5 (5.3) | 39.1 (4.9) | 40 (5.1)
  Physical Health: Post-intervention, One week: number analyzed (Participants) | 77 | 77 | 75 | 76
  Physical Health: Post-intervention, One week | 40.2 (4.7) | 39.6 (5.5) | 39.6 (4.6) | 40.5 (5.0)
  Physical Health: Post-intervention, six months: number analyzed (Participants) | 77 | 77 | 75 | 75
  Physical Health: Post-intervention, six months | 38.7 (5.2) | 38.7 (5.6) | 39.2 (4.5) | 40.0 (5.1)
  Physical Health 12 months post-intervention: number analyzed (Participants) | 77 | 76 | 74 | 75
  Physical Health 12 months post-intervention | 39.5 (5.3) | 39.1 (6.2) | 38.9 (5.1) | 39.3 (5.1)
  Mental Health: Baseline | 50.8 (7.4) | 52.3 (7.9) | 51.8 (8.0) | 52.9 (8.1)
  Mental Health: Post-intervention, One week: number analyzed (Participants) | 77 | 77 | 75 | 76
  Mental Health: Post-intervention, One week | 53.1 (7.1) | 52.4 (7.9) | 52.2 (8.3) | 53.8 (8.0)
  Mental Health: Post-intervention, Six months: number analyzed (Participants) | 77 | 77 | 75 | 75
  Mental Health: Post-intervention, Six months | 51.4 (7.0) | 50.6 (8.2) | 51.7 (7.4) | 52.8 (8.4)
  Mental Health: Post-intervention, Twelve months: number analyzed (Participants) | 77 | 76 | 74 | 75
  Mental Health: Post-intervention, Twelve months | 51.1 (7.4) | 50.3 (8.3) | 50.3 (7.4) | 49.9 (8.3)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Otago,PAM, Inter+Intra Strategies: Condition 4:
  1. Otago Exercise Program (OEP) adapted for delivery to small groups. In total, this protocol includes 5 flexibility movements, 5 leg-strengthening movements, and 12 balance-challenging movements. The number intensity and duration (dosages) are individualized according to preference and ability. OEP movements are gradually progressed across the 8-week intervention.
  2. A physical activity monitor (PAM) (Fitbit Charge 2) with initial orientation and ongoing support.
  3. Interpersonal behavior change strategies including peer-to-peer sharing and learning about using activities in everyday routines as prompts for movement, identifying and problem solving environmental barriers to physical activity, ways to increase social support for physical activity, and friendly social comparison of experiences performing OEP movements and home and other locations of choice, staying motivated to practice OEP movements long-term.
  4. Intrapersonal behavior change strategies including to develop physical activity related goals and action plans, self-assess goal attainment and action plan implementation-adjust accordingly, identify and problem solve personal barriers to physical activity, develop a habit of one or more OEP movement
Arm/Group | Otago+PAM+Health / Wellness Topics | Otago + PAM + Interpersonal Strategies | Otago, PAM, Intrapersonal Strategies | Otago,PAM, Inter+Intra Strategies
All-Cause Mortality (participants affected / at risk) | 1/77 | 2/76 | 1/74 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/76 | 0/74 | 2/75
Other Adverse Events (participants affected / at risk) | 2/77 | 7/76 | 3/74 | 3/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Otago+PAM+Health / Wellness Topics (N=77) | Otago + PAM + Interpersonal Strategies (N=76) | Otago, PAM, Intrapersonal Strategies (N=74) | Otago,PAM, Inter+Intra Strategies (N=75)
cancer (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stroke (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Otago+PAM+Health / Wellness Topics (N=77) | Otago + PAM + Interpersonal Strategies (N=76) | Otago, PAM, Intrapersonal Strategies (N=74) | Otago,PAM, Inter+Intra Strategies (N=75)
Pain (General disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Fall (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
fracture (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Polymyalgia rheumatica--unrelated (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cancer (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
lung illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hyponatremia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT03326141/Prot_SAP_002.pdf
  • Informed Consent Form (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT03326141/ICF_003.pdf